CLINICAL TRIAL: NCT00730119
Title: Evaluation Of The GE Monitor Product Line
Status: Withdrawn | Type: Observational
Why Stopped: Terminated due to lack of enrollment at target sites
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: CS 327
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Non-invasive Blood Pressure; Temperature; SpO2; Respiration; ECG
Keywords: Non-invasive Blood Pressure (NIBP); GE Monitor; Temperature; SpO2; Respiration, ECG
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Neonates: Subjects ages birth to 30 days
- Infants: Subjects aged >30 days to 2 years
- Adults: Subjects aged 18 years of age or older

SUMMARY:
This investigation is a multi-center study that will demonstrate that the GE Monitor meets equivalency and/or accuracy and/or performance criteria. This investigation will compare the test device(s) to itself, or one of the reference parameters, or a combination of parameters, including NIBP, temperature, SpO2, respirations, and ECG.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from subject and/or guardian
* Ability to maintain proper placement of cuff and/or probe and/or sensor
* Presence of atrial fibrillation or other irregular heart rhythm (when applicable)
* Ability to single or dual monitor NIBP, ECG, and/or SpO2, whether or not already being monitored for any or all of these parameters (SuperSTAT development study only)

Exclusion Criteria:

* Any subject deemed too unstable, by clinician's discretion, or for another reason deemed unacceptable for study by the clinician
* Known dysrhythmias (when applicable)
* Known disease state or medical condition that A) compromises circulation to the extremity, B) compromises musculo-skeletal integrity, or C) otherwise contraindicates use of a NIBP cuff and/or SpO2 sensor on an extremity or ECG patches on skin
* Vigorous exercise prior to participating in the study
* Excessive movement or excitability causing false values or no determinations
* Known allergy to latex when latex products will be in contact with subject
* Subjects who have eaten, drank, smoked or chewed gum in the preceding half hour (temperature parameter only)
* Nasal/septal defects, cold and/or allergies that would not allow the subject to breathe through their nose (temperature parameter only)
* Subjects with whom flammable anesthetics will be used.
* Adult/pediatric subjects,(greater than 1 year of age) who, at the clinician's discretion, could not tolerate approximately 12, but no more than 25 blood pressures on each extremity
* Pediatric/neonatal subjects,(less than 1 year of age) who, at the clinician's discretion, could not tolerate approximately 10, but no more than 12 blood pressures on each extremity
* Presence of pacemaker which makes the atrial fibrillation rhythm indistinguishable
* Subject's limb circumference is outside of the manufacturer's recommended cuff range
* Subject has Korotkoff sounds that persist to nearly zero (when applicable)

Min Age: 1 Minute | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All populations (neonatal, pediatrics, and adults).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2001-10 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
This investigation will compare values from the test device(s) to itself, or one of the reference parameters, or a combination of parameters, including NIBP, temperature, SpO2, respirations, and ECG. | unlimited

CONTACTS AND LOCATIONS:
Overall Officials: Jean D Sesing, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Tampa, Florida, United States